CLINICAL TRIAL: NCT04099186
Title: Evaluation of Safety and Efficacy of Hydro-mechanical Defragmentation of High Risk Pulmonary Embolism With Contraindications to Thrombolytic Therapy
Brief Title: Hydro-mechanical Defragmentation of Pulmonary Embolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman khairy Mohamed, assisstant professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMDPE
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: non randomized case control trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: inclusion in each arm was made by pulmonary embolism response team not by the investigators . also at level of follow up assessment was done by blinded investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydro-mechanical pulmonary embolism fragmentation (Experimental): Those patients will undergo catheter directed fragmentation followed by injection of 100 ml of heparinized saline via power injector
  Interventions: Procedure: catheter directed hydro-mechanical fragmentation of pulmonary embolism
- thrombolytic treated arm (No Intervention): patients with high risk and intermediate high risk PE who received thrombolysis as only treatment modality

INTERVENTIONS:
Procedure: catheter directed hydro-mechanical fragmentation of pulmonary embolism — A(6)F multipurpose catheter will be advanced over a guide wire under fluoroscopic guidance and used to measure right heart and pulmonary artery pressures, then mechanical catheter fragmentation will be done using a pigtail catheter. The catheter will be quickly spun manually so as to fragment the central thrombus and establish initial flow into pulmonary artery , then 200 ml saline will be injected via power injector to aid fragmentation of thrombus
  Arms: hydro-mechanical pulmonary embolism fragmentation

SUMMARY:
Evaluating the safety and outcomes of hydro-mechanical defragmentation of high risk pulmonary embolism with contraindication for thrombolytic therapy

DETAILED DESCRIPTION:
In high risk pulmonary embolism , the main aim of therapy is to rapidly recanalize the affected pulmonary arteries with thrombolysis or embolectomy; to decrease right ventricular afterload and reverse right ventricular failure and shock, prevent chronic thromboembolic pulmonary hypertension , and decrease the recurrence risk.

The first-line treatment in patients with acute high risk pulmonary embolism presenting with persistent hypotension and/or cardiogenic shock is intravenous thrombolytic therapy. However a significant proportion of patients may not be a candidate for Intravenous thrombolysis because of major contraindications. An alternative option in patients with absolute contraindications or has failed intravenous thrombolysis is surgical embolectomy , but the number of experienced tertiary care centers that can do emergency surgical embolectomy are limited.

Percutaneous catheter mechanical fragmentation of proximal pulmonary arterial clots followed by injection of 200 ml saline at high pressure using power injector can be used as an alternative to intravenous thrombolytic therapy and surgical embolectomy because of their ability to rapidly recanalize occluded pulmonary blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angiographically confirmed acute high risk pulmonary embolism with shock index >1.
* Pulmonary arterial occlusion with >50% involvement of the central (main and/or lobar) pulmonary , and pulmonary hypertension (mean pulmonary artery pressure >25 mmHg)
* Patients with high risk pulmonary embolism who cannot receive fibrinolysis
* Patients with acute intermediate-high risk pulmonary embolism with adverse prognosis (new hemodynamic instability, worsening respiratory failure, severe RV (right ventricle) dysfunction, or major myocardial necrosis)

Exclusion Criteria:

* Patients with echocardiographically confirmed right sided thrombi.
* Patients with low-risk pulmonary embolism or intermediate-low risk acute pulmonary embolism with minor RV dysfunction, minor myocardial necrosis, and no clinical worsening
* Anaphylactic reaction to contrast media.
* Acute renal failure or severe chronic non-dialysis dependent kidney disease.
* Uncooperative patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  measure the estimates of deaths in the 30 days after pulmonary embolism diagnosis

SECONDARY OUTCOMES:
oxygen saturation | 24 hours
  oxygen saturation will be measured by arterial blood gases analysis at first admission and compared with measurements the following second, eighth, and 24th hours of the intervention
Changes in blood pressure | 24 hours
  systolic and diastolic blood pressure will be measured at first admission and compared with measurements the following second, eighth, and 24th hours of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Uflacker R. Interventional therapy for pulmonary embolism. J Vasc Interv Radiol. 2001 Feb;12(2):147-64. doi: 10.1016/s1051-0443(07)61821-1. PMID 11265879
- [Background] Engelberger RP, Kucher N. Reperfusion Treatment for Acute Pulmonary Embolism. Hamostaseologie. 2018 May;38(2):98-105. doi: 10.1055/s-0038-1641717. Epub 2018 May 29. PMID 29843174
- [Background] Kuo WT, Banerjee A, Kim PS, DeMarco FJ Jr, Levy JR, Facchini FR, Unver K, Bertini MJ, Sista AK, Hall MJ, Rosenberg JK, De Gregorio MA. Pulmonary Embolism Response to Fragmentation, Embolectomy, and Catheter Thrombolysis (PERFECT): Initial Results From a Prospective Multicenter Registry. Chest. 2015 Sep;148(3):667-673. doi: 10.1378/chest.15-0119. PMID 25856269
- [Background] Mohan B, Chhabra ST, Aslam N, Wander GS, Sood NK, Verma S, Mehra AK, Sharma S. Mechanical breakdown and thrombolysis in subacute massive pulmonary embolism: A prospective trial. World J Cardiol. 2013 May 26;5(5):141-7. doi: 10.4330/wjc.v5.i5.141. PMID 23710301
- [Background] Dilektasli AG, Demirdogen Cetinoglu E, Acet NA, Erdogan C, Ursavas A, Ozkaya G, Coskun F, Karadag M, Ege E. Catheter-Directed Therapy in Acute Pulmonary Embolism with Right Ventricular Dysfunction: A Promising Modality to Provide Early Hemodynamic Recovery. Med Sci Monit. 2016 Apr 15;22:1265-73. doi: 10.12659/msm.897617. PMID 27081754
- [Derived] Hassan AKM, Ahmed H, Ahmed Y, Elfadl AA, Omar A. Efficacy and safety of hydro-mechanical defragmentation in intermediate- and high-risk pulmonary embolism. Egypt Heart J. 2021 Sep 25;73(1):84. doi: 10.1186/s43044-021-00204-2. PMID 34564780